CLINICAL TRIAL: NCT04456959
Title: A Retrospective Chart Review of UK Patients With Relapsed/Refractory Acute Lymphoblastic Leukaemia Treated With Inotuzumab Ozogamicin, a Real World Research Study
Brief Title: InO - A Retrospective Study of UK Patients With Leukaemia
Acronym: InO
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001222
Record Dates: First submitted 2020-06-08; First posted 2020-07-07 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult R/R ALL patients who have received InO: Relapsed/refractory ALL patients who are 18 years and over and initiated InO between 1st of June 2016 and date of data collection (to be confirmed). They will have accessed InO treatment via NHS commissioning, via the CUP, or via private purchase and will have at least 3 months follow up from the index date unless death occurs within that time.
  Interventions: Drug: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin — Inotuzumab ozogamicin is an antibody-drug conjugate (ADC) composed of a recombinant humanised IgG4 kappa CD22-directed monoclonal antibody (produced in Chinese hamster ovary cells by recombinant DNA technology) that is covalently linked to N-acetyl-gamma-calicheamicin dimethylhydrazide.
  Other Names: CMC-544

SUMMARY:
The purpose of this study is to describe the demographics and clinical characteristics, treatment pathway, and effectiveness and safety of inotuzumab ozogamicin in patients with relapsed/refractory B-cell acute lymphoblastic leukaemia treated with inotuzumab ozogamicin in the real-world.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory ALL.
* Patients who initiated InO between 1st of June 2016 and date of data collection.
* Patients who accessed InO treatment via NHS commissioning, via the CUP, or via private purchase.
* Patient aged ≥18 years old at initiation of InO treatment

Exclusion Criteria:

* Patients initiated on treatment with InO at a different hospital than the ones selected in this study.
* Patients with <3 months of follow-up since index date, unless death occurs <3 months from index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed/refractory Acute Lymphoblastic Leukemia who are aged 18 and over and initiated Inotuzumab Ozogamicin between 1st of June 2016 and date of data collection and received treatment via NHS commissioning, via the Compassionate Use Programme, or via private purchase.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United Kingdom (4):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - University College London Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust of Fulham Road, London
  - Taunton and Somerset NHS Foundation Trust of Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who initiated treatment with inotuzumab ozogamicin (InO) for relapsed/refractory B-cell acute lymphoblastic leukemia (ALL), in real world settings as a part of routine clinical care, between June 2016 and January 2021, were included. Data of these participants, were retrieved from hospital records and observed in this retrospective, observational study for approximately 1 year duration.
Groups:
- Inotuzumab Ozogamicin (InO): Participants with relapsed/refractory B-cell ALL, were treated with InO in real world settings as part of routine clinical care, between June 2016 to January 2021. Data of these participants were studied for approximately 1 year in this study.
Period: Overall Study
Arm/Group | Inotuzumab Ozogamicin (InO)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised of medical records extracted for the purpose of the study from all eligible participants who were included in the study.
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Time from ALL Diagnosis to Index Date [Mean (Standard Deviation); unit: Years] — Here, time from ALL diagnosis to index date was reported. Index date: date of initiation of the first cycle of InO.
  Years | 2.6 (5.3)
Number of Participants According to Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS is used to measure quality of life of oncology participants with scores ranging from 0 to 5;where 0= fully active, able to carry on all pre-disease performance without restriction;1= restricted in physically strenuous activity, ambulatory, able to carry out light or sedentary work;2= ambulatory, capable of all self-care, unable to carry out any work activity, up greater than (>)50 percent (%) of waking hours;3= capable of only limited self-care, confined to bed or chair >50% of waking hours;4= completely disabled, cannot carry on any self-care, totally confined to bed or chair;5= dead.
  Participants
    0 | 5
    1 | 4
    Not recorded | 19
Number of Participants According to Their Phase of Disease at Index Date [Count of Participants; unit: Participants] — Here, number of participants are classified according to phase of ALL disease: complete remission (CR), 1st relapse, 2nd relapse, 3rd relapse, 4th or greater relapse. Remission = either the reduction or disappearance of the signs and symptoms of a disease. Relapse = return of a disease or the signs and symptoms of a disease after a period of improvement. Index date: date of initiation of the first cycle of InO.
  Participants
    First relapse | 21
    Second relapse | 6
    Third relapse | 1
    Fourth or greater relapse | 0
    CR | 0
Number of Participants According to History of Liver Disease Recorded for Prior to Index Date Period [Count of Participants; unit: Participants] — Here, number of participants are classified according to their history of liver disease prior to index date, as 1) No = no previous liver disease history, 2) Yes = previous liver disease history and 3) Not know. Prior to index date period: time post ALL diagnosis to index date. Index date: date of initiation of the first cycle of InO.
  Participants
    No | 22
    Not known | 5
    Yes | 1
Percentage of Positive Cell Blasts (CD22 expression test) [Mean (Standard Deviation); unit: Percentage of cells] — Population: Here number analyzed signifies participants evaluable for this baseline characteristic.
  Percentage of cells
    number analyzed (Participants) | 8
    (all) | 49.6 (29.6)
Number of Participants According to ALL Mutation Types [Count of Participants; unit: Participants] — Here, number of participants were classified per ALL mutation type.
  Participants
    (1;19)(q23;p13) | 1
    BCR-ABL | 4
    Complex karyotype | 1
    Cytogenetics failed | 1
    ETV6 Rearrangement | 1
    Gain 18 centromere | 1
    Gain part of chr 5 | 1
    Not Known | 16
    Relapse with clonal evolution | 1
    t(8:14) | 1
Blood Platelet Counts [Mean (Standard Deviation); unit: cells*10^9 per liter] | 95.9 (76.2)
Blood Absolute Neutrophil Counts [Mean (Standard Deviation); unit: cells*10^9 per liter] — Population: Here number analyzed signifies participants evaluable for this baseline characteristic.
  cells*10^9 per liter
    number analyzed (Participants) | 18
    (all) | 4.1 (6.5)
Blood Alanine Aminotransferase (ALT) Levels [Mean (Standard Deviation); unit: International units per liter (IU/L)] | 37.9 (35.3)
Blood Aspartate Aminotransferase (AST) Levels [Mean (Standard Deviation); unit: International units per liter] — Population: Here number analyzed signifies participants evaluable for this baseline characteristic.
  International units per liter
    number analyzed (Participants) | 2
    (all) | 29 (2.8)
Blood Bilirubin Levels [Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)] — Population: Here number analyzed signifies participants evaluable for this baseline characteristic.
  Milligrams per deciliter (mg/dL)
    number analyzed (Participants) | 25
    (all) | 0.6 (0.4)
Blood Albumin Levels [Mean (Standard Deviation); unit: Grams per deciliter (g/dL)] | 3.6 (0.7)
Blood Gamma Glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: Units per liter (U/L)] — Population: Here number analyzed signifies participants evaluable for this baseline characteristic.
  Units per liter (U/L)
    number analyzed (Participants) | 5
    (all) | 74.8 (82.7)
Blood Alkaline Phosphatase (ALP) Levels [Mean (Standard Deviation); unit: International units per liter] — Population: Here number analyzed signifies participants evaluable for this characteristic.
  International units per liter
    number analyzed (Participants) | 27
    (all) | 112.7 (95.1)
Number of Participants According to Number of ALL Relapses Recorded for Prior to Index Date Period [Count of Participants; unit: Participants] — Here, number of participants are classified according to number of relapses of ALL relapse prior to index date. Prior to index date period: time post ALL diagnosis to index date. Index date: date of initiation of the first cycle of InO.
  Participants
    1 | 21
    2 | 5
    3 | 1
    Not known | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received First Line Chemotherapy According to National Trial or Treatment Guideline
Description: In this outcome measure, number of participants who were treated with the first-line chemotherapy during anytime between initial diagnosis of ALL and InO initiation, were reported.
Time Frame: Anytime between initial diagnosis of ALL and InO initiation, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  At least one line of prior chemotherapy recorded | 27
  Not recorded | 1

2. Primary Outcome: Number of Participants According to Number of Lines of Salvage Therapy
Description: In this outcome measure, number of participants according to number of lines of salvage therapy anytime between initial diagnosis of ALL and InO initiation, were reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  1 | 6
  2 | 1
  No salvage therapy | 21

3. Primary Outcome: Number of Participants According to Prior Hematopoietic Stem Cell Transplant (HSCT)
Description: In this outcome measure, number of participants, who were treated with hematopoietic stem cell transplant (HSCT) before initiation of InO, were reported.
Time Frame: Anytime between initial diagnosis of ALL and InO initiation, during data identification period from June 2016 to January 2021 (approximately 4.5 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  At least one line of prior HSCT recorded | 10
  No prior HSCT | 15
  Not recorded | 3

4. Primary Outcome: Number of Participants According to Type of Conditioning Regimen for Each HSCT
Description: In this outcome measure, number of participants were classified according to different type of conditioning regimen for each HSCT (high-dose intensity myeloablative, reduced-intensity/non-myeloablative), were reported.
Time Frame: as for outcome 1
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who had at least 1 line of prior HSCT recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 10
Participants
  High-dose intensity myeloablative | 7
  Not known | 1
  Reduced intensity/ non-myeloablative | 2

5. Primary Outcome: Number of Participants Who Were Treated Previously With Blinatumomab
Description: In this outcome measure, number of participants who were previously treated with blinatumomab, were reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Prior treatment with blinatumomab | 4
  No prior treatment with Blinatumomab | 24

6. Primary Outcome: Number of Participants Treated With Chimeric Antigen Receptor (CAR) T-Cell Therapies
Description: In this outcome measure, number of participants treated with chimeric antigen receptor (CAR) T-cell therapies before initiation of InO, were reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Participants with prior CAR T-Cell therapy | 0
  Participants with no prior CAR T-Cell therapy | 18
  Not recorded | 10

7. Secondary Outcome: Total Duration of Treatment With Inotuzumab Ozogamicin
Description: In this outcome measure, total duration of InO treatment was reported.
Time Frame: From InO initiation date to date of end of treatment, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Days | 71.4 (52.4)

8. Secondary Outcome: Number of Participants According to Number of Inotuzumab Ozogamicin Treatment Cycles
Description: In this outcome measure, number of participants were classified according to total number of InO treatment cycles received.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Received Total of 1 Cycle | 6
  Received Total of 2 Cycles | 13
  Received Total of 3 Cycles | 5
  Received Total of 4 Cycles | 2
  Received Total of 5 Cycles | 0
  Received Total of 6 Cycles | 2

9. Secondary Outcome: Number of Participants According to Interrupted Inotuzumab Ozogamicin Treatment Cycles
Description: In this outcome measure, number of participants were classified according to number of interrupted cycles of InO treatment.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  0 Cycle Interrupted | 20
  1 Cycle Interrupted | 7
  2 Cycle Interrupted | 1

10. Secondary Outcome: Number of Participants According to Reasons for Inotuzumab Ozogamicin Treatment Interruption
Description: In this outcome measure, number of participants, were reported according to reasons of interruption in respective Cycles.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, 'number analyzed' signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Cycle 1: Cycle was not Interrupted | 24
  Cycle1: Interrupted Due to Death: number analyzed (Participants) | 4
  Cycle1: Interrupted Due to Death | 1
  Cycle 1:Interrupted Due to Liver toxicity Treatment Related Adverse Events (TRAEs): number analyzed (Participants) | 4
  Cycle 1:Interrupted Due to Liver toxicity Treatment Related Adverse Events (TRAEs) | 1
  Cycle 1: Interrupted Due to Neutropenia and Severe Constipation: number analyzed (Participants) | 4
  Cycle 1: Interrupted Due to Neutropenia and Severe Constipation | 1
  Cycle 1: Interrupted Due to SARS-CoV 2 infection: number analyzed (Participants) | 4
  Cycle 1: Interrupted Due to SARS-CoV 2 infection | 1
  Cycle 2: Cycle was not Interrupted: number analyzed (Participants) | 22
  Cycle 2: Cycle was not Interrupted | 19
  Cycle 2: Interrupted Due to High Fever, Rigors, Vomiting, Hypotension: number analyzed (Participants) | 3
  Cycle 2: Interrupted Due to High Fever, Rigors, Vomiting, Hypotension | 1
  Cycle 2: Interrupted Due to Liver Toxicity TRAE(s): number analyzed (Participants) | 3
  Cycle 2: Interrupted Due to Liver Toxicity TRAE(s) | 1
  Cycle 2: Interrupted Due to Nausea, Poor oral intake, Neutropenic Sepsis: number analyzed (Participants) | 3
  Cycle 2: Interrupted Due to Nausea, Poor oral intake, Neutropenic Sepsis | 1
  Cycle 3: Cycle was not Interrupted: number analyzed (Participants) | 9
  Cycle 3: Cycle was not Interrupted | 7
  Cycle 3: Interrupted Due to Infection in Peripherally Inserted Central Catheter: number analyzed (Participants) | 2
  Cycle 3: Interrupted Due to Infection in Peripherally Inserted Central Catheter | 1
  Cycle 3: Interrupted Due to Transferred to Another Hospital: number analyzed (Participants) | 2
  Cycle 3: Interrupted Due to Transferred to Another Hospital | 1

11. Secondary Outcome: Number of Participants According to Prescribed Inotuzumab Ozogamicin Doses
Description: In this outcome measure, number of participants according to prescribed starting InO dose, were reported.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, 'number analyzed' signifies participants evaluable for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Cycle 1: 0.8 milligram per meter square (mg/m^2) | 1
  Cycle 1: 1.8 mg/m^2 | 27
  Cycle 2: 1.0 mg/m2: number analyzed (Participants) | 22
  Cycle 2: 1.0 mg/m2 | 1
  Cycle 2: 1.2 mg/m^2: number analyzed (Participants) | 22
  Cycle 2: 1.2 mg/m^2 | 1
  Cycle 2: 1.5 mg/m^2: number analyzed (Participants) | 22
  Cycle 2: 1.5 mg/m^2 | 9
  Cycle 2: 1.8 mg/m^2: number analyzed (Participants) | 22
  Cycle 2: 1.8 mg/m^2 | 11
  Cycle 3: 1.5 mg/m^2: number analyzed (Participants) | 9
  Cycle 3: 1.5 mg/m^2 | 4
  Cycle 3: 1.8 mg/m^2: number analyzed (Participants) | 9
  Cycle 3: 1.8 mg/m^2 | 5
  Cycle 4: 0.5 mg/m^2: number analyzed (Participants) | 4
  Cycle 4: 0.5 mg/m^2 | 1
  Cycle 4: 1.5 mg/m^2: number analyzed (Participants) | 4
  Cycle 4: 1.5 mg/m^2 | 3
  Cycle 5: 1.5 mg/m^2: number analyzed (Participants) | 2
  Cycle 5: 1.5 mg/m^2 | 2
  Cycle 6: 1.5 mg/m^2: number analyzed (Participants) | 2
  Cycle 6: 1.5 mg/m^2 | 2

12. Secondary Outcome: Number of Participants Classified on the Basis of Any Modifications in Inotuzumab Ozogamicin Dose
Description: In this outcome measure, number of participants were classified as following: 1) with no dose modification and 2) no data recorded.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, number analyzed signifies participants evaluable for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Cycle 1: Participants with no dose modification | 26
  Cycle 1: No data recorded | 2
  Cycle 2: number analyzed (Participants) | 22
  Cycle 2: Participants with no dose modification | 20
  Cycle 2: No data recorded | 2
  Cycle 3: number analyzed (Participants) | 9
  Cycle 3: Participants with no dose modification | 7
  Cycle 3: No data recorded | 2
  Cycle 4: number analyzed (Participants) | 4
  Cycle 4: Participants with no dose modification | 3
  Cycle 4: No data recorded | 1
  Cycle 5: number analyzed (Participants) | 2
  Cycle 5: Participants with no dose modification | 2
  Cycle 5: No data recorded | 0
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6: Participants with no dose modification | 2
  Cycle 6: No data recorded | 0

13. Secondary Outcome: Number of Participants Who Were Treated With Concomitant Azole Antifungal Therapy
Description: In this outcome measure, number of participants who were treated with concomitant azole antifungal therapy along with InO treatment were reported.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Not Treated With Concomitant Azole Antifungal Therapy | 26
  Treated With Concomitant Azole Antifungal Therapy | 2

14. Secondary Outcome: Duration of Concomitant Azole Antifungal Therapy
Description: In this outcome measure, time/duration between start date and end date of concomitant azole antifungal, was reported.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here 'overall number of participants analyzed' signifies participants evaluable for this outcome measure and were treated with concomitant azole antifungal therapy.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Days | 20 (1.4)

15. Secondary Outcome: Number of Participants Who Achieved Complete Remission (CR) by the End of InO Treatment
Description: CR was defined as documented in medical records or (if unavailable in the records) as less than (<) 5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets greater than or equal to [>=] 100*10^9 cells per liter [/L] and absolute neutrophil counts [ANC] >=1*10^9 cells/L) and resolution of any extramedullary disease.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants | 15

16. Secondary Outcome: Number of Participants Who Achieved CR With Incomplete Hematological Recovery (CRi) by the End of InO Treatment
Description: CRi was defined as documented in medical records or (if unavailable in the records) <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100* 10^9 cells/L and ANC <1*10^9 cells/L) and resolution of any extramedullary disease.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants | 5

17. Secondary Outcome: Number of Participants With CR/CRi by the End of InO Treatment
Description: In this outcome, number of participants who achieved CR/CRi at the end of InO treatment are reported. CR was defined as documented in medical records or as <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets >=100*10^9 cells/L and ANC >=1*10^9 cells/L) and resolution of any extramedullary disease. CRi was defined as documented in medical records or <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100*10^9 cells/L and ANC <1*10^9 cells/L) and resolution of any extramedullary disease.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants | 20

18. Secondary Outcome: Median Time to CR/CRi
Description: CR was defined as documented in medical records or as <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets >=100*10^9 cells/L and ANC >=1*10^9 cells/L) and resolution of any extramedullary disease. CRi was defined as documented in medical records or <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100*10^9 cells/L and ANC <1*10^9 cells/L) and resolution of any extramedullary disease.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here 'overall number of participants analyzed' signifies participants evaluable for this outcome measure with CR/CRi.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 20
Months | 1.7 [1.6 to 4.3]

19. Secondary Outcome: Number of Participants Who Achieved Negative Minimal Residual Disease (MRD) Among Those Who Had CR/CRi
Description: Negative MRD was defined as documented in medical records or (if unavailable in the records) as leukemic cells comprising <1*10^-4 (<0.01%) of bone marrow nucleated cells. This outcome measure was analyzed in participants with CR/CRi. CR was defined as documented in medical records or as <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets >=100*10^9 cells/L and ANC >=1*10^9 cells/L) and resolution of any extramedullary disease. CRi was defined as documented in medical records or <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100*10^9 cells/L and ANC <1*10^9 cells/L) and resolution of any extramedullary disease.
Time Frame: as for outcome 7
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 20
Participants | 14

20. Secondary Outcome: Number of Participants Who Achieved Negative MRD Classified Per InO Cycles
Description: Negative MRD (among those who had CR/CRi) was defined as documented in medical records or (if unavailable in the records) as leukemic cells comprising <1*10^-4 (<0.01%) of bone marrow nucleated cells. CR was defined as documented in medical records or as <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets >=100*10^9 cells/L and ANC >=1*10^9 cells/L) and resolution of any extramedullary disease. CRi was defined as documented in medical records or <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100*10^9 cells/L and ANC <1*10^9 cells/L) and resolution of any extramedullary disease.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here 'overall number of participants analyzed' signifies participants evaluable for this outcome measure with negative MRD.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 14
Participants
  1 | 1
  2 | 7
  3 and above | 6

21. Secondary Outcome: Number of Participants Who Survived at 3, 6 and 12 Months Post InO Treatment Initiation
Description: In this outcome measure, number of participants who survived 3, 6, and 12 post InO treatment, were reported.
Time Frame: At 3, 6, and 12 months post InO initiation date, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  3 months | 25
  6 months | 19
  12 months | 13

22. Secondary Outcome: Number of Participants Classified According to Their Cause of Death
Description: In this outcome measure, number of participants according to their cause of death were reported.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 19
Participants
  Acute Lymphoblastic Leukaemia | 15
  Pneumonia | 1
  SAR COV 2 | 1
  Subarachnoid/Intraparenchymal Hemorrhage Stroke | 1
  Veno-Occlusive Disease | 1

23. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the index date to the date of death. Participants were censored at date of latest visit at the time of data collection. Kaplan-Meier method was used for OS analysis.
Time Frame: InO initiation date to death due to any cause or last visit at time of data collection, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Months | 11.7 [6.3 to NA] — Upper limit of 95% CI could not be estimated because there were insufficient number of participants with event.

24. Secondary Outcome: Percentage of Participants Who Were Relapse-free at 3, 6 and 12 Months Post InO Treatment Initiation
Description: Relapse free survival: the time from the start of treatment to earliest date of the following events: death, progressive disease (including objective progression, relapse from CR/CRi, treatment discontinuation due to global deterioration of health status), and start of new induction therapy or post-therapy HSCT without achieving CR/CRi; as documented in medical records. CR: documented in medical records or as <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets >=100*10^9/L and ANC >=1*10^9/L) and resolution of any extramedullary disease. CRi: documented in medical records or <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100*10^9/L and ANC <1*10^9/L) and resolution of any extramedullary disease. Progressive disease (PD): a doubling of peripheral blasts with an absolute increase of >5*10^9 cells/L.
Time Frame: At 3, 6, and 12 months from InO initiation date, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Percentage of participants
  3 months | 82.1 [69.1 to 97.6]
  6 months | 60.7 [45.1 to 81.8]
  12 months | 39.3 [24.8 to 62.3]

25. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined as the time from the start of treatment to earliest date of the following events: death, PD (including objective progression, relapse from CR/CRi, treatment discontinuation due to global deterioration of health status), and start of new induction therapy or post-therapy HSCT without achieving CR/CRi; as documented in medical records. CR was defined as documented in medical records or as <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets >=100*10^9 cells /L and ANC >=1*10^9 cells/L) and resolution of any extramedullary disease. CRi was defined as documented in medical records or <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100*10^9 cells/L and ANC <1*10^9 cells/L) and resolution of any extramedullary disease. PD: a doubling of peripheral blasts with an absolute increase of >5*10^9 cells/L.
Time Frame: From InO initiation date to death or progressive disease, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Months | 8.86 [4.93 to NA] — Upper limit of 95% CI was not estimable due insufficient number of participants with event.

26. Secondary Outcome: Time to Non-relapse Mortality (NRM)
Description: NRM was defined as the time from the date of follow-up HSCT until death due to any cause without disease progression or relapse.
Time Frame: Post InO treatment from date of follow up HSCT to death, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, "Overall number of Participants" signifies evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 9
Months | 12.69 [5.88 to NA] — Upper limit of 95% CI was not estimable due insufficient number of participants with event.

27. Secondary Outcome: Number of Participants According to Types of Therapies Post Inotuzumab Ozogamicin Treatment
Description: In this outcome measure, number of participants according to therapies they initiated post InO treatment were reported. One participant could have more than 1 type of therapies.
Time Frame: Post InO treatment, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Chemotherapy | 16
  HSCT | 9
  CAR-T cell therapy | 8

28. Secondary Outcome: Number of Participants Who Achieved CR, CRi, Progressive Disease and Stable Disease With Different Types of Post Inotuzumab Ozogamicin Treatments
Description: CR was defined as documented in medical records or as <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, full recovery of peripheral blood counts (platelets >=100*10^9 cells/L and ANC >=1*10^9 cells/L) and resolution of any extramedullary disease. CRi was defined as documented in medical records or <5% blasts in the bone marrow and the absence of peripheral blood leukemic blasts, incomplete recovery of peripheral blood counts (platelets <100*10^9 cells/L and ANC <1*10^9 cells/L) and resolution of any extramedullary disease. PD was defined as a doubling of peripheral blasts with an absolute increase of >5*10^9 cells/L. Stable disease was defined as increase of peripheral blasts with an absolute increase not >50%.
Time Frame: as for outcome 27
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, 'number analyzed' signifies participants evaluable for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  HSCT: CR: number analyzed (Participants) | 9
  HSCT: CR | 5
  HSCT: CRi: number analyzed (Participants) | 9
  HSCT: CRi | 3
  HSCT: Not Known: number analyzed (Participants) | 9
  HSCT: Not Known | 1
  CAR-T cell therapy: CR: number analyzed (Participants) | 8
  CAR-T cell therapy: CR | 5
  CAR-T cell therapy: CRi: number analyzed (Participants) | 8
  CAR-T cell therapy: CRi | 1
  CAR-T cell therapy: PD: number analyzed (Participants) | 8
  CAR-T cell therapy: PD | 1
  CAR-T cell therapy: Not Known: number analyzed (Participants) | 8
  CAR-T cell therapy: Not Known | 2
  Blinatumomab: CR: number analyzed (Participants) | 8
  Blinatumomab: CR | 2
  Blinatumomab: Not Recorded: number analyzed (Participants) | 8
  Blinatumomab: Not Recorded | 2
  Blinatumomab: PD: number analyzed (Participants) | 8
  Blinatumomab: PD | 3
  Blinatumomab: SD: number analyzed (Participants) | 8
  Blinatumomab: SD | 1
  Other Chemotherapy: CR: number analyzed (Participants) | 16
  Other Chemotherapy: CR | 3
  Other Chemotherapy: CRi: number analyzed (Participants) | 16
  Other Chemotherapy: CRi | 4
  Other Chemotherapy: Missing: number analyzed (Participants) | 16
  Other Chemotherapy: Missing | 1
  Other Chemotherapy: Not Recorded: number analyzed (Participants) | 16
  Other Chemotherapy: Not Recorded | 11
  Other Chemotherapy: PD: number analyzed (Participants) | 16
  Other Chemotherapy: PD | 4
  Other Chemotherapy: SD: number analyzed (Participants) | 16
  Other Chemotherapy: SD | 1

29. Secondary Outcome: Number of Participants Who Survived Post InO Blinatumomab Treatment
Description: In this outcome measure, number of participants who survived at completion of InO treatment were reported.
Time Frame: as for outcome 27
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 8
Participants | 8

30. Secondary Outcome: Number of Participants Who Experienced a Documented Diagnosis of Veno-occlusive Disease (VOD)/Sinusoidal Obstruction Syndrome (SOS) Post InO Treatment
Description: VOD, also called SOS, happens when the small blood vessels that lead into the liver and are inside the liver become blocked.
Time Frame: as for outcome 27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Participants With VOD/SOS | 2
  Participants Not With VOD/SOS | 26

31. Secondary Outcome: Number of Participants According to Type of Treatments Received for Documented Diagnoses of Veno-occlusive Disease (VOD)/Sinusoidal Obstruction Syndrome (SOS)
Description: as for outcome 30
Time Frame: as for outcome 27
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure with VOD/SOS.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Participants
  Spironolactone | 1
  Ursodeoxycholic Acid | 1

32. Secondary Outcome: Number of Participants Who Survived Following Treatment For Documented Diagnoses of Veno-occlusive Disease (VOD)/Sinusoidal Obstruction Syndrome (SOS)
Description: as for outcome 30
Time Frame: as for outcome 27
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Participants | 1

33. Secondary Outcome: Number of Participants With Interrupted InO Treatment Due to VOD/SOS
Description: as for outcome 30
Time Frame: as for outcome 27
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Participants | 2

34. Secondary Outcome: Number of Participants With Moderate Severity VOD/SOS
Description: as for outcome 30
Time Frame: Post InO Treatment, during data identification period from June 2016 to January 2021 (approximately 4.5 years); from the data collected and observed retrospectively over approximately 12 months of this study
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Participants | 2

35. Secondary Outcome: Number of Participants Who Experienced Grade 3 and Grade 4 (Lung/Cardiac/Kidney/Liver) Treatment Related Adverse Event (TRAE) Following Inotuzumab Ozogamicin Initiation
Description: Adverse event (AE) was defined as any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 3 were severe events. Grade 4 were life-threatening events. Information for grades was recorded as per participants' medical records.
Time Frame: as for outcome 7
Population: Safety analysis set (SAS) included the medical records extracted for the purpose of the study from all eligible participants who were included in the study and had at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants
  Grade 3 | 1
  Grade 4 | 1

36. Secondary Outcome: Number of Participants According to Types of Treatments Received for Grade3/4 TRAE Following Inotuzumab Ozogamicin Initiation
Description: AE was defined as any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 3 were severe events. Grade 4 were life-threatening events. Information for grades was recorded as per participants' medical records.
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure with Grade 3 or 4 TRAE.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 2
Participants
  Antibiotics/ Intensive Therapy Unit | 1
  High dose septrin + Caspofungi | 1

37. Secondary Outcome: Number of Participants With Liver Dysfunction Following Inotuzumab Ozogamicin Initiation
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 28
Participants | 1

38. Secondary Outcome: Number of Participants With Peripheral Blood Blast Counts Measurement Prior to Post InO HSCT
Time Frame: Prior to post InO HSCT, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 5
Participants | 0

39. Secondary Outcome: Number of Participants With Significant Risk Factors for VOD/SOS
Description: In this outcome measure, participants with significant risk factor for VOD/ SOS occurrence were reported. VOD, also called SOS, happens when the small blood vessels that lead into the liver and are inside the liver become blocked
Time Frame: as for outcome 7
Population: FAS included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and number analyzed signifies participants evaluable for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin (InO)
Number analyzed (Participants) | 9
Participants
  Number of alkylating agents:1: number analyzed (Participants) | 8
  Number of alkylating agents:1: Experienced VOD/SOS: Yes | 1
  Number of alkylating agents:1: Experienced VOD/SOS: No | 7
  Number of alkylating agents: 3: number analyzed (Participants) | 1
  Number of alkylating agents: 3: Experienced VOD/SOS: Yes | 0
  Number of alkylating agents: 3: Experienced VOD/SOS: No | 1
  Busulfan-containing regimen: Experienced VOD/SOS: Yes | 1
  Busulfan-containing regimen: Experienced VOD/SOS: No | 8
  Last bilirubin concentration prior to follow-up HSCT: > upper limit normal (ULN): number analyzed (Participants) | 1
  Last bilirubin concentration prior to follow-up HSCT: > upper limit normal (ULN): Experienced VOD/SOS: Yes | 0
  Last bilirubin concentration prior to follow-up HSCT: > upper limit normal (ULN): Experienced VOD/SOS: No | 1
  Last bilirubin concentration prior to follow-up HSCT: <ULN: number analyzed (Participants) | 7
  Last bilirubin concentration prior to follow-up HSCT: <ULN: Experienced VOD/SOS: Yes | 1
  Last bilirubin concentration prior to follow-up HSCT: <ULN: Experienced VOD/SOS: No | 6
  Last bilirubin concentration prior to follow-up HSCT: Missing: number analyzed (Participants) | 1
  Last bilirubin concentration prior to follow-up HSCT: Missing: Experienced VOD/SOS: Yes | 0
  Last bilirubin concentration prior to follow-up HSCT: Missing: Experienced VOD/SOS: No | 1
  Age: <55 years: number analyzed (Participants) | 8
  Age: <55 years: Experienced VOD/SOS: Yes | 1
  Age: <55 years: Experienced VOD/SOS: No | 7
  Age: >55 years: number analyzed (Participants) | 1
  Age: >55 years: Experienced VOD/SOS: Yes | 0
  Age: >55 years: Experienced VOD/SOS: No | 1
  Last ALT concentration prior to follow-up HSCT: less than or equal to (≤)1.5 ULN: number analyzed (Participants) | 8
  Last ALT concentration prior to follow-up HSCT: less than or equal to (≤)1.5 ULN: Experienced VOD/SOS: Yes | 1
  Last ALT concentration prior to follow-up HSCT: less than or equal to (≤)1.5 ULN: Experienced VOD/SOS: No | 7
  Last ALT concentration prior to follow-up HSCT: Missing: number analyzed (Participants) | 1
  Last ALT concentration prior to follow-up HSCT: Missing: Experienced VOD/SOS: Yes | 0
  Last ALT concentration prior to follow-up HSCT: Missing: Experienced VOD/SOS: No | 1
  Last AST concentration prior to follow-up HSCT: ≤1.5 ULN: number analyzed (Participants) | 1
  Last AST concentration prior to follow-up HSCT: ≤1.5 ULN: Experienced VOD/SOS: Yes | 0
  Last AST concentration prior to follow-up HSCT: ≤1.5 ULN: Experienced VOD/SOS: No | 1
  Last AST concentration prior to follow-up HSCT: Missing: number analyzed (Participants) | 8
  Last AST concentration prior to follow-up HSCT: Missing: Experienced VOD/SOS: Yes | 1
  Last AST concentration prior to follow-up HSCT: Missing: Experienced VOD/SOS: No | 7

ADVERSE EVENTS:
Time Frame: From InO initiation date to date of end of treatment, during data identification period from June 2016 to January 2021 (approximately 4.7 years); retrieved data was analyzed during 12 months of this observational study
Description: Same event may appear as both an AE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AEs were reported as per participants' medical records. There was no specific medical dictionary.
Arm/Group | Inotuzumab Ozogamicin (InO)
All-Cause Mortality (participants affected / at risk) | 19/28
Serious Adverse Events (participants affected / at risk) | 2/28
Other Adverse Events (participants affected / at risk) | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (InO) (N=28)
Lung (General disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (InO) (N=28)
Veno-occlusive Disease (VOD)/Sinusoidal Obstruction Syndrome (SOS) (General disorders) | 2
Liver (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT04456959/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT04456959/SAP_001.pdf